CLINICAL TRIAL: NCT00454142
Title: A Phase 2 Study of GW786034 (Pazopanib) in Asian Patients With Recurrent/Metastatic Nasopharyngeal Carcinoma
Brief Title: Pazopanib Hydrochloride in Treating Patients With Stage IV or Recurrent Nasopharyngeal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00197; NCI-2009-00197 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000537520 (Registry Identifier: NCI); CTRG-NP05/25/06 (Other: Cancer Therapeutics Research Group (CTRG)); NCC-06-01 (Other: National Cancer Centre); 7623 (Other: CTEP)
Record Dates: First submitted 2007-03-27; First posted 2007-03-30 (Estimated); Results first posted 2015-12-17 (Estimated); Last update posted 2015-12-17 (Estimated); Status verified 2012-01

CONDITIONS: Recurrent Lymphoepithelioma of the Nasopharynx; Recurrent Squamous Cell Carcinoma of the Nasopharynx; Stage IV Lymphoepithelioma of the Nasopharynx; Stage IV Squamous Cell Carcinoma of the Nasopharynx
MeSH Terms: interventions — pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (pazopanib hydrochloride) (Experimental): Patients receive pazopanib hydrochloride PO QD on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Pharmacological study will be done on Day 1 and Day 28. Computed tomography will be done at baseline and day 28.
  Interventions: Drug: pazopanib hydrochloride; Other: pharmacological study; Procedure: computed tomography

INTERVENTIONS:
Drug: pazopanib hydrochloride — Given PO
  Other Names: GW786034B; Votrient
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Procedure: computed tomography — Correlative studies
  Other Names: tomography, computed

SUMMARY:
This phase II trial studies the side effects and how well pazopanib hydrochloride works in treating patients with stage IV or recurrent nasopharyngeal cancer. Pazopanib hydrochloride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the efficacy of pazopanib hydrochloride in patients with stage IV or recurrent nasopharyngeal carcinoma.

II. Determine the progression-free survival of patients treated with this drug. III. Determine the toxicity of this drug in these patients. IV. Determine the effect of this drug on angiogenesis inhibition using dynamic contrast-enhanced computed tomography (CT) scan.

V. Determine the pharmacokinetic profile of this drug in these patients. VI. Correlate the effect of this drug on angiogenesis inhibition with the clinical benefit rate and pharmacokinetics.

OUTLINE:

Patients receive pazopanib hydrochloride orally (PO) once daily (QD) on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically for up to 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed nasopharyngeal carcinoma, meeting the following criteria:

  * World Health Organization (WHO) type II-III disease
  * Stage IV or recurrent disease
* Must have failed at least 1 prior line of chemotherapy for metastatic or recurrent disease
* Measurable disease, defined as >= 1 unidimensionally measurable lesion >= 20 mm by conventional techniques OR >= 10 mm by spiral CT scan
* No known brain metastases
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-2 or Karnofsky PS 70-100%
* Life expectancy > 3 months
* WBC >= 3,000/mm³
* Absolute neutrophil count >= 1,500/mm³
* Platelet count >= 100,000/mm³
* Bilirubin normal
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 times upper limit of normal (ULN)
* Creatinine normal OR creatinine clearance >= 60 mL/min
* Proteinuria =< 1+ on 2 consecutive dipsticks taken >= 1 week apart
* Prothrombin time (PT), international normalized ratio (INR), and partial thromboplastin time (PTT) =< 1.2 times ULN
* Systolic blood pressure (BP) =< 140 mm Hg and diastolic BP =< 90 mm Hg

  * Initiation or adjustment of BP medication allowed provided the average of 3 BP readings are < 140/90 mm Hg prior to study entry
* No history of allergic reaction attributed to compounds of similar chemical or biological composition to pazopanib hydrochloride or to other study agents
* No abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 28 days
* No cerebrovascular accident within the past 6 months
* No history of any of the following diseases within the past 12 weeks:

  * Myocardial infarction
  * Cardiac arrhythmia
  * Admission for unstable angina
  * Cardiac angioplasty or stenting
  * Venous thrombosis
* No New York Heart Association (NYHA) class III-IV heart failure

  * Patients with a history of NYHA class II heart failure are eligible provided they are asymptomatic on treatment
* No significant electrocardiogram (ECG) abnormalities, including QTc prolongation (i.e., QTc >= 500 msec)
* No serious or non-healing wound, ulcer, or bone fracture
* No condition that would impair the ability to swallow and retain pazopanib hydrochloride, including any of the following:

  * Gastrointestinal tract disease resulting in an inability to take oral medication
  * Requirement for IV alimentation
  * Prior surgical procedures affecting absorption
  * Active peptic ulcer disease
* No concurrent uncontrolled illness including, but not limited to, the following:

  * Coagulopathy
  * Ongoing or active infection
  * Psychiatric illness or social situation that would preclude study compliance
* No known allergy to CT contrast agents
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin C) and recovered
* More than 4 weeks since prior radiotherapy
* At least 4 weeks since prior surgery
* No prior antiangiogenesis therapy
* No other concurrent investigational agents
* No other concurrent anticancer therapy
* No concurrent medications or substances known to affect or with the potential to affect the activity or pharmacokinetics of pazopanib hydrochloride, as determined by the Principal Investigator
* No concurrent medications that have the potential to interact with the cytochrome P450 (CYP) isoenzymes CYP2C9 and CYP3A4
* No concurrent therapeutic warfarin

  * Low molecular weight heparin or prophylactic low-dose warfarin allowed
* No concurrent antiretroviral therapy for human immunodeficiency virus (HIV)-positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2007-08; Primary Completion 2010-04 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wan Teck Lim, Principal Investigator — National Cancer Centre
Locations (3):
- Singapore (3):
  - Cancer Therapeutics Research Group, Singapore
  - National University Hospital, Singapore
  - National Cancer Centre, Singapore

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were screened and enrolled from 2 sites in Singapore, 27 were enrolled from National Cancer Centre Singapore and 6 were enrolled from National University Hospital.
Pre-assignment Details: Once a subject signed the informed consent form, the required screening procedures would be performed.Eligible subjects would undergo 2 times of DCE-CT scan before study drug administration.
Groups:
- Treatment (Tyrosine Kinase Inhibitor): Patients receive pazopanib hydrochloride PO QD on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  computed tomography : Correlative studies
  pharmacological study : Correlative studies
  pazopanib hydrochloride : Given PO
Period: Overall Study
Arm/Group | Treatment (Tyrosine Kinase Inhibitor)
Started | 33
Completed | 32
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Tyrosine Kinase Inhibitor)
Number analyzed (Participants) | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 31
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 23
Region of Enrollment [Number; unit: participants]
  Singapore | 33

OUTCOME MEASURES:

1. Secondary Outcome: Response Rate (PR)
Description: Per response evaluation criteria in solid tumors (RECIST v1.0) and assessed by MRI or CT: Partial response (PR), >=30% decrease in the sum of the longest diameter of target lesions and non-PD (PD: progressive disease) of non-target lesions.
Time Frame: 12 weeks of treatment
Measure: Number; unit: percentage of participants
Groups:
- Treatment (Pazopanib Hydrochloride): Patients receive pazopanib hydrochloride PO QD on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  pazopanib hydrochloride: Given PO
  pharmacological study: Correlative studies
  computed tomography: Correlative studies
Arm/Group | Treatment (Pazopanib Hydrochloride)
Number analyzed (Participants) | 33
percentage of participants | 6.1

2. Secondary Outcome: Progression-free Survival
Description: Progression will be evaluated in this study using the new international criteria proposed by RECIST Committee. The sample proportion and associated 95% confidence interval will be reported.
Time Frame: From the date of enrollment to the date of first documented progression or death, whichever occurs first, or to the date when the patient was last known to be alive, up to 3 years.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Tyrosine Kinase Inhibitor)
Number analyzed (Participants) | 33
months | 4.4 [3.9 to 5.8]

3. Primary Outcome: Clinical Benefit Rate
Description: Clinical benefit rate (CBR) as defined by Response Evaluation Criteria in Solid Tumors (RECIST ver 1.0) and assessed by CT or MRI. CBR includes 1) Complete response (CR): disappearance of all lesions; 2) partial response (PR): >=30% decrease in the sum of the longest diameter of target lesions and 3) stable disease (SD): non-PR and non progressive disease.
Time Frame: 12 weeks of treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Treatment (Tyrosine Kinase Inhibitor): Patients receive pazopanib hydrochloride PO daily (QD) on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  computed tomography : Correlative studies
  pharmacological study : Correlative studies
  pazopanib hydrochloride : Given PO
Arm/Group | Treatment (Tyrosine Kinase Inhibitor)
Number analyzed (Participants) | 33
percentage of participants | 54.5 [38.0 to 70.2]

4. Secondary Outcome: Overall Survival
Time Frame: From date of enrollment to the study to the date of death from any cause or to the date when the patient was last known to be alive, up to 3 years.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Pazopanib Hydrochloride)
Number analyzed (Participants) | 33
months | 10.8 [8.6 to 21.8]

5. Secondary Outcome: Toxicity Profile: Percentage of Participants With Significant (Grade 3/4) Related Adverse Event (AE)
Description: The frequencies of grade 3/4 related toxicities were recorded among all participants, and the percentage of participants who experienced significant AEs were reported.
Time Frame: From the time of first treatment with pazopanib hydrochloride to up to 30days after completion of treatment
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (Tyrosine Kinase Inhibitor)
Number analyzed (Participants) | 33
percentage of participants | 48

6. Secondary Outcome: Pharmacodynamic Study: Tumor Blood Flow at Baseline
Description: Dynamic-contrast enhanced computed tomography (DCE-CT) was performed at baseline and Day 28, tumor blood flow was measured.19 of 33 patients had evaluable DCE-CT data.
Time Frame: Pretreatment
Measure: Mean (Standard Deviation); unit: ml/100ml/min
Arm/Group | Treatment (Pazopanib Hydrochloride)
Number analyzed (Participants) | 19
ml/100ml/min | 52.2 (13.6)

7. Secondary Outcome: Pharmacodynamic Study: Tumor Blood Flow on Day 28
Description: DCE-CT was performed on Day 28 and tumor blood flow was measured. 19 of 33 patients had evaluable DCE-CT data.
Time Frame: 28 days post treatment
Measure: Mean (Standard Deviation); unit: ml/100ml/min
Arm/Group | Treatment (Pazopanib Hydrochloride)
Number analyzed (Participants) | 19
ml/100ml/min | 35.7 (18.5)

8. Secondary Outcome: Pharmacokinetic Study: Percentage of Participants With Trough Concentration at Steady State (Day 28) Above 15 µg/mL
Description: Pazopanib pharmacokinetic parameters were estimated on Day 1 and Day 28 (steady state). Trough concentration of pazopanib was measured on Day 28 with blood sampling at zero (pre dose), 0.5 hr, 1, 2, 3, 4, 5, 6, 8 and 24 hrs after Day 28 dose.
Time Frame: Day 28 of treatment
Population: Patients (total 26) with both Day 1 and Day 28 pharmacokinetic parameters were included.The trough concentration of pazopanib on Day 28 was observed to be above 15ug/ml in approximately 92% of patients at steady state.
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (Pazopanib Hydrochloride)
Number analyzed (Participants) | 26
percentage of participants | 92

9. Secondary Outcome: Pharmacokinetic Study: AUC0-24h/Dose on Day 1
Description: AUC 0-24h/dose were measured on day 1 for 26 evaluable participants. Blood sampling is done at zero (pre-dose), 0.5 hr, 1, 2, 3, 4, 5, 6 and 8 hrs after the first dose.
Time Frame: Day 1 of treatment
Measure: Median (Full Range); unit: hr*ng/mL/mg
Arm/Group | Treatment (Pazopanib Hydrochloride)
Number analyzed (Participants) | 26
hr*ng/mL/mg | 836.23 [165.73 to 1869.21]

10. Secondary Outcome: Pharmacokinetic Study: Area Under Curve (AUC) 0-24h/Dose on Day 28
Description: AUC 0-24h/dose were measured on day 28 for 26 evaluable participants. Blood sampling was done at zero (pre dose), 0.5 hr, 1, 2, 3, 4, 5, 6, 8 and 24 hrs after day 28 dose.
Time Frame: Day 28 of treatment
Measure: Median (Full Range); unit: hr*ng/mL/mg
Arm/Group | Treatment (Pazopanib Hydrochloride)
Number analyzed (Participants) | 26
hr*ng/mL/mg | 1192.35 [82.96 to 4345.95]

11. Secondary Outcome: Pharmacokinetic Study: Volume of Distribution (Vd/F/Dose) on Day 1
Description: Volume of distribution (Vd/F/dose) were measured on day 1 for 26 evaluable participants. Blood sampling was done at zero (pre dose), 0.5 hr, 1, 2, 3, 4, 5, 6, 8 hrs after first dose.
Time Frame: Day 1 of treatment
Measure: Median (Full Range); unit: mL/mg
Arm/Group | Treatment (Pazopanib Hydrochloride)
Number analyzed (Participants) | 26
mL/mg | 18.09 [8.34 to 79.02]

12. Secondary Outcome: Pharmacokinetic Study: Volume of Distribution at Steady State (Vss/F/Dose) on Day 28
Description: Volume of distribution at steady state (Vss/F/Dose) were measured on day 28 for 26 evaluable participants. Blood sampling was done at zero (pre dose), 0.5 hr, 1, 2, 3, 4, 5, 6, 8 and 24 hrs after day 28 dose.
Time Frame: Day 28 of treatment
Measure: Median (Full Range); unit: mL/mg
Arm/Group | Treatment (Pazopanib Hydrochloride)
Number analyzed (Participants) | 26
mL/mg | 80.23 [16.58 to 1601.70]

ADVERSE EVENTS:
Time Frame: From the time of first treatment with pazopanib hydrochloride to up to 1 month after completion of treatment.
Arm/Group | Treatment (Tyrosine Kinase Inhibitor)
Serious Adverse Events (participants affected / at risk) | 10/33
Other Adverse Events (participants affected / at risk) | 11/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Tyrosine Kinase Inhibitor) (N=33)
infection (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pericardial effusion (Cardiac disorders) | 1 (1)
Hemorrhage (Blood and lymphatic system disorders) | 3 (3)
Hyperbilirubin (Hepatobiliary disorders) | 1 (1)
Pain (Nervous system disorders) | 1 (1)
Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Tyrosine Kinase Inhibitor) (N=33)
Anorexia (Gastrointestinal disorders) | 3 (3)
Dehydration (General disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Fatigue (General disorders) | 5 (5)
Hand-foot-skin reaction (Skin and subcutaneous tissue disorders) | 5 (5)
Hypertension (Cardiac disorders) | 1 (1)
hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Lethargy (General disorders) | 1 (1)
Neutropenic fever (Blood and lymphatic system disorders) | 1 (1)
Proteinuria (Metabolism and nutrition disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less